CLINICAL TRIAL: NCT04479540
Title: Assessment of the Risk of Pulmonary Embolism and Coagulation Profile in Patients With SARS Coronavirus (COV-2) Lung Disease
Brief Title: Assessment of the Risk of Pulmonary Embolism and Coagulation Profile in Patients With COVID-19 Lung Disease
Acronym: COVIDEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Hospital Ambroise Paré Paris (Other); University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020_0058
Record Dates: First submitted 2020-07-06; First posted 2020-07-21 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Pneumonia, Viral
Keywords: SARS COV-2; pulmonary embolism; acute respiratory distress syndrome; coagulation disorders; venous thromboembolic disease
MeSH Terms: conditions — Pneumonia, Viral; Pulmonary Embolism; Respiratory Distress Syndrome; Hemostatic Disorders

STUDY DESIGN:
Intervention Model Description: Determination of incidence of occurrence of pulmonary embolism in hospitalized patients with SARS-CoV-2 pneumonitis, first by performing systematic thoracic angiography scanner in all hospitalized patients and then to explore hemostasis profile
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hospitalized SARS Cov-2 (Experimental): Hospitalized patients diagnosed with SARS Cov-2 infection
  Interventions: Radiation: Angiography scanner

INTERVENTIONS:
Radiation: Angiography scanner — systematic thoracic angiography scanner to diagnose pulmonary embolism and additional blood sample (hemostasis exploration)

SUMMARY:
The current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic is complicated by pneumonia (15 to 20% of cases) requiring hospitalization with oxygen therapy. Almost 20 to 25% of hospitalized patients require intensive care and resuscitation; half die.

The main cause of death is acute respiratory distress syndrome (ARDS). However, some deaths have been linked to pulmonary embolism (PE).

Recognition of PE is important because there is specific treatment to limit its own mortality. The identification of biological parameters of hemostasis predictive of thromboembolic disease is crucial in these patients.

To evaluate the frequency of PE in the patients having to be hospitalized is to practice of a systematic thoracic angiography scanner in the patients having no contra-indication for its realization, as well as during hospitalization in patients deteriorating without any other obvious cause.

The thromboembolic events and disturbances of the coagulation system described in patients with SARS-CoV-2 pneumonitis suggest that this viral infection is associated with an increase in the activation of coagulation contributing to the occurrence of thrombosis and especially from PE.

DETAILED DESCRIPTION:
The current severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) pandemic is complicated by pneumonia (15 to 20% of cases) requiring hospitalization with oxygen therapy. Almost 20 to 25% of hospitalized patients require intensive care and resuscitation; half die.

On April 3, 2020, in France, 59,105 confirmed cases have been identified. 6,305 people are hospitalized in intensive care and 4,503 patients died.

The main cause of death is acute respiratory distress syndrome (ARDS). However, some deaths have been linked to pulmonary embolism (PE). Very little data is available in the medical literature regarding PE during this infection.

Recognition of PE is important because there is specific treatment to limit its own mortality. The identification of biological parameters of hemostasis predictive of thromboembolic disease is crucial in these patients who are difficult to mobilize.

The diagnostic difficulties with traditional means, the seriousness and the ignorance of a PE make it necessary to evaluate the frequency of it in the patients having to be hospitalized by the practice of a systematic thoracic angiography scanner in the patients having no contra-indication for its realization, as well as during hospitalization in patients deteriorating without any other obvious cause.

The thromboembolic events and disturbances of the coagulation system described in patients with SARS-CoV-2 pneumonitis suggest that this viral infection is associated with an increase in the activation of coagulation contributing to the occurrence of thrombosis and especially from PE.

The main objective of this work is therefore to determine the incidence of the occurrence of PE in patients with hospitalized SARS-CoV-2 pneumonitis by performing systematic thoracic angiography scanner in all hospitalized patients.

The secondary objective is to study the coagulation and fibrinolysis profile in these patients and to assess endothelial activation in order to better understand the physio-pathological mechanism behind PE and to determine if one of the parameters studied could be an indicator of PE risk.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Any patient who consults in the emergency room, COVID+ with hospitalization criteria (dyspnea or desaturation ≤ 95% or chest pain or hemoptysis), including those who have already performed a CT angiogram upon arrival at the hospital.
* Positive polymerase chain reaction (PCR) of coronavirus disease or compatible clinical signs associated with suggestive radiological criteria

  * Fever
  * Cough
  * Myalgia
  * Asthenia
  * Loss of taste/ Anosmia
* signed informed consent before any study procedure
* patients affiliated to an appropriate health insurance system

Exclusion Criteria:

* Pregnancy in progress
* Patient not having a microbiological diagnosis of SARS Coronavirus (COV-2) infection or whose symptoms are not suggestive
* < 18 years
* Be deprived of liberty or under guardianship
* Patient with contra-indication to thoracic angiography scanner:

  * State of shock
  * Creatinine clearance < 30 mL/mn in Chronic Kidney Disease (CKD)
  * history of anaphylactic shock or angioedema with iodinated contrast media
  * uncontrolled cardiac decompensation
* Patient with contra-indication to contrast media (Iomeron350®, Visipaque®):

  * History of immediate major or delayed skin reaction to the injection of a contrast medium
  * Hypersensitivity to the active substance or to any of the excipients
  * overt thyrotoxicosis

Patients with renal insufficiency and / or patients with allergy to iodinated contrast products may be included if they can perform a scintigraphy (the pulmonary scintigraphy being the alternative diagnostic to the CT angiography for renal insufficiency and / or allergy to iodinated contrast products).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Rate of patients with pulmonary embolism | up to Day 12
  Rate of patients with pulmonary embolism diagnosed by thoracic angiography scanner

SECONDARY OUTCOMES:
Prothrombin level measurement | up to Day 12
  Measure of prothrombin level to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
activated partial thromboplastin time measurement | up to Day 12
  Measure of activated partial thromboplastin time to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Fibrinogen measurement | up to Day 12
  Measure of fibrinogen to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
D-dimers measurement | up to Day 12
  Measure of D-dimers to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Protein C measurement | up to Day 12
  Measure of Protein C to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Willebrand antigen measurement | up to Day 12
  Measure of Willebrand antigen to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Soluble tissue factor measurement | up to Day 12
  Measure of Soluble tissue factor to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Soluble thrombomodulin measurement | up to Day 12
  Measure of soluble thrombomodulin to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
E-selectin measurement | up to Day 12
  Measure of E-selectin to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Thrombin-antithrombin complex measurement | up to Day 12
  Measure of thrombin-antithrombin complex to assess hemostasis parameters of patients with SARS-COV-2pneumonitis during hospitalization
Assessment of clot formation curve | Day 1
  Assessment of clot formation curve by Thrombodynamics® to identify ones predictive of the onset of Pulmonary Embolism or a poor prognosis
Assessment of thrombin generation | Day 1
  Assessment of thrombin generation by Thrombodynamics® to identify ones predictive of the onset of Pulmonary Embolism or a poor prognosis
Assessment of fibrinolysis | Day 1
  Assessment of fibrinolysis by Thrombodynamics® to identify ones predictive of the onset of Pulmonary Embolism or a poor prognosis
Mortality | Day 30
  Determine patient mortality

CONTACTS AND LOCATIONS:
Overall Officials: Colas TCHERAKIAN, MD, Principal Investigator — Foch HOSPITAL
Locations (1):
- Hôpital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No